CLINICAL TRIAL: NCT04223609
Title: Non-intrusive Detection of Temporary Neurologic Impairment By Opioids
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gaurav N. Pradhan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-004883
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Oxycodone, Then Placebo (Experimental): Participants first receive initial dose of oxycodone 5 mg tablet followed by a 30-minute rest period to allow for onset of medication effect. This rest period will be followed by a standardized set of oculomotor testing for 40 minutes. After the initial testing, a second dose of oxycodone 5 mg tablet will be administered followed by a 30-minute rest period to allow for the onset of the second dose. The second rest period will be followed by a second round of standardized oculomotor testing for 40 minutes. Participants will then return approximately 4 to 6 days to repeat the standardized oculomotor testing with placebo.
  Interventions: Drug: Oxycodone; Drug: Placebo; Device: EyeLink 1000 Plus; Diagnostic Test: Oculo-Cognitive Addition test (OCAT); Device: VT3mini - Eye Tracking Technology for OEMs
- Placebo, Then Oxycodone (Experimental): Participants first receive initial dose of placebo 5 mg tablet followed by a 30-minute rest period to allow for onset of medication effect. This rest period will be followed by a set of standardized oculomotor testing for 40 minutes. After the initial testing, a second dose of placebo 5 mg tablet will be administered followed by a 30-minute rest period to allow for the onset of the second dose. The second rest period will be followed by a second round of standardized oculomotor testing for 40 minutes. Participants will then return approximately 4 to 6 days to repeat the standardized oculomotor testing with oxycodone.
  Interventions: Drug: Oxycodone; Drug: Placebo; Device: EyeLink 1000 Plus; Diagnostic Test: Oculo-Cognitive Addition test (OCAT); Device: VT3mini - Eye Tracking Technology for OEMs

INTERVENTIONS:
Drug: Oxycodone — 5 mg tablet
  Other Names: Oxycodone Immediate Release
Drug: Placebo — Oxycodone-matched placebo tablet
Device: EyeLink 1000 Plus — Non-invasive video-based eye tracking system
  Other Names: EyeLink
Diagnostic Test: Oculo-Cognitive Addition test (OCAT) — Subject will have to look for numbers on a screen and add these numbers together. OCAT will be presented on a computer screen with attached eye tracking device at the bottom part.
Device: VT3mini - Eye Tracking Technology for OEMs — Non-invasive eye-tracking device
  Other Names: EyeTech

SUMMARY:
Research is being conducted to better understand the physiologic effects (relating to the action of a drug when taken by a healthy person) of opioid use on oculomotor (relating to the motion of the eye) dynamics and to identify the presence of characteristics consistent with a specific drug or class of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to consent to participate themselves
* Be healthy male or non-pregnant female
* Must be able to attend in-person sessions at the Mayo Aerospace Medicine and Vestibular Research Laboratory in Scottsdale, AZ.
* Have not used opioids during the preceding 30 days
* Prior use of opioids for pain management

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Women who are not practicing an effective form of contraception (condoms, IUD, birth control pill, diaphragm),
* Past or current history of drug or substance use.
* Significant ocular disorder.
* Positive drug test for marijuana, opioids, methamphetamines, cocaine, PCP or other controlled substances.
* History of use of psychoactive drugs within the past 30 days.
* Subjects with a history of cardiopulmonary disease including but not limited to congestive heart failure, obstructive sleep apnea, restrictive lung disease, COPD, moderate to severe asthma and oxygen dependency.
* Subjects currently taking sedatives (including benzodiazepines), muscle relaxants or disassociatives.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Pradhan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxycodone, Then Placebo | Placebo, Then Oxycodone
Started | 6 | 8
Completed | 6 | 6
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Missed last visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone, Then Placebo | Placebo, Then Oxycodone | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.3) | 32.6 (8.2) | 31.2 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Oculo-Cognitive Addition Test (OCAT) Completion Time
Description: Time it takes participants to complete the OCAT measured in seconds.
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Oxycodone: Participants who received initial dose of oxycodone 5 mg tablet followed by a 30-minute rest period to allow for onset of medication effect. This rest period will be followed by a standardized set of oculomotor testing for 40 minutes. After the initial testing, a second dose of oxycodone 5 mg tablet will be administered followed by a 30-minute rest period to allow for the onset of the second dose. The second rest period will be followed by a second round of standardized oculomotor testing for 40 minutes.
- Placebo: Participants who received initial dose of placebo 5 mg tablet followed by a 30-minute rest period to allow for onset of medication effect. This rest period will be followed by a set of standardized oculomotor testing for 40 minutes. After the initial testing, a second dose of placebo 5 mg tablet will be administered followed by a 30-minute rest period to allow for the onset of the second dose. The second rest period will be followed by a second round of standardized oculomotor testing for 40 minutes.
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
seconds
  Baseline | 57.22 (10.23) | 57.22 (10.23)
  Approx. 30 minutes after initial 5 mg dose | 59.56 (12.01) | 58.18 (10.15)
  Approx. 30 minutes after second 5 mg dose | 56.12 (11.81) | 54.47 (12.66)

2. Primary Outcome: Saccadic Latency
Description: measured in seconds
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
seconds
  Baseline | 0.40 (0.07) | 0.40 (0.07)
  Approx. 30 minutes after initial 5 mg dose | 0.45 (0.13) | 0.38 (0.08)
  Approx. 30 minutes after second 5 mg dose | 0.38 (0.08) | 0.38 (0.10)

3. Primary Outcome: Fixation Time - Low Cognitive Workload
Description: measure in milliseconds
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
milliseconds
  Baseline | 1079.82 (187.66) | 1079.82 (187.66)
  Approx. 30 minutes after initial 5 mg dose | 1145.60 (239.89) | 1198.86 (204.36)
  Approx. 30 minutes after second 5 mg dose | 1132.70 (285.69) | 1073.96 (260.28)

4. Primary Outcome: Fixation Time - Medium Cognitive Workload
Description: measure in milliseconds
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
milliseconds
  Baseline | 1316.45 (239.58) | 1316.45 (239.58)
  Approx. 30 minutes after initial 5 mg dose | 1347.90 (236.69) | 1381.20 (286.50)
  Approx. 30 minutes after second 5 mg dose | 1249.38 (329.62) | 1264.03 (346.36)

5. Primary Outcome: Fixation Time - High Cognitive Workload
Description: measure in milliseconds
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
milliseconds
  Baseline | 1572.63 (303.23) | 1572.63 (303.23)
  Approx. 30 minutes after initial 5 mg dose | 1644.75 (344.26) | 1641.86 (345.10)
  Approx. 30 minutes after second 5 mg dose | 1564.34 (324.77) | 1528.17 (419.64)

6. Primary Outcome: Diagonal Saccadic Velocity
Description: measured in deg/s
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: deg/s
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
deg/s
  Baseline | 284.81 (31.32) | 284.81 (31.32)
  Approx. 30 minutes after initial 5 mg dose | 293.82 (36.48) | 277.44 (44.99)
  Approx. 30 minutes after second 5 mg dose | 281.42 (31.95) | 285.74 (25.84)

7. Primary Outcome: Horizontal Saccadic Velocity
Description: measured in deg/s
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: deg/s
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
deg/s
  Baseline | 302.93 (28.54) | 302.93 (28.54)
  Approx. 30 minutes after initial 5 mg dose | 288.52 (25.29) | 283.77 (27.21)
  Approx. 30 minutes after second 5 mg dose | 289.74 (32.77) | 286.66 (23.57)

8. Primary Outcome: Vertical Saccadic Velocity
Description: measured in deg/s
Time Frame: Baseline, post initial dose (approximately 30 minutes) and post second dose (approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: deg/s
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 13
deg/s
  Baseline | 298.52 (38.30) | 298.52 (38.30)
  Approx. 30 minutes after initial 5 mg dose | 274.51 (28.73) | 272.93 (48.12)
  Approx. 30 minutes after second 5 mg dose | 309.83 (126.58) | 276.21 (27.38)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately one week on all participants.
Arm/Group | Oxycodone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 1/13 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone (N=13) | Placebo (N=14)
Nausea and dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04223609/Prot_SAP_000.pdf